CLINICAL TRIAL: NCT06802354
Title: Application of Gaseous Ozone in the Surgical Extraction of Impacted Mandibular Third Molars: Impact on the Incidence of Postoperative Complications and Healing Processes
Brief Title: Efficacy of Ozone Therapy in Reducing Complications Following Impacted Mandibular Third-molar Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jelena Krunic (Other)
Responsible Party: Sponsor-Investigator, Jelena Krunic, Associate Professor, University of East Sarajevo
Organization: University of East Sarajevo (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-2-9; 19.032/961-110/23 (Other Grant/Funding Number: Ministry of Scientific and Technological Development and Higher Education, Republic of Srpska)
Record Dates: First submitted 2024-12-16; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Impacted Mandibular Third Molar Extraction
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Intervention Model Description: The study is a 'split-mouth' randomized clinical controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone therapy (Experimental): After the surgical extraction of the impacted mandibular third molar, gaseous ozone will be applied at the extraction site. Ozone will be reapplied 3 days after the intervention, according to the manufacturer's recommendation for wound treatment following tooth extraction.
  Interventions: Drug: Ozone
- Sham Comparator (Sham Comparator): After the surgical extraction of the impacted mandibular third molar, a sham ozone therapy will be applied at the extraction site. The sham ozone therapy will also be reapplied 3 days after the surgical intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozone — In Ozone group, ozone will be applied at the site of the extraction wound for 30 seconds after the surgical extraction of the third molar, according to the manufacturer's recommendation for wound treatment following tooth extraction.
  Arms: Ozone therapy
Drug: Placebo — In the control group, a sham ozone therapy will be applied at the site of the extraction wound for 30 seconds after the surgical extraction of the third molar .
  Arms: Sham Comparator

SUMMARY:
The goal of this clinical trial is to learn if use of ozone works to treat complications after impacted mandibular third molar surgery. It will also learn does ozone has positive effect on wound healing and quality of life.

The main questions it aims to answer are:

* Does ozone reduce incidence of postoperative compliactions such as pain, swelling or reduced mouth opening after impacted mandibular third molar surgery?
* Does ozone improve wound healing after impacted mandibular third molar surgery?
* Does ozone have positive effect on quality of life after impacted mandibular third molar surgery?

Participants will:

* Receive ozone after impacted mandibular third molar surgery.
* Visit the clinic 1st, 3rd, and 7th days after the intervention for checkups and tests.
* Keep a diary of their symptoms.

DETAILED DESCRIPTION:
The aims of this study were: (i) to determine the effects of gaseous ozone on pain, swelling, and trismus and healing process measured by cytokine levels, and (ii) to measure patient quality of life after impacted mandibular third molar surgery.

All participants included in the study will be informed about the aims and expected outcomes of the research, the sample collection procedure, and will sign an informed consent form. All participants will be treated according to the principles of good clinical practice and in accordance with the Helsinki Declaration. The Ethics Committee of the Faculty of Medicine provide study approval.

The surgical procedure for each patient will be performed using a standardized surgical technique in two clinical visits (one side per visit).

The surgical area will be disinfected. To ensure pain relief during the procedure, local anesthesia will be applied using blocks of the inferior alveolar and buccal nerves. After elevating the flap, osteotomy will be performed with a carbide drill using an air drill and continuous irrigation with saline solution. Depending on the morphology of the tooth, the third molar will either be extracted or the crown will be separated from the roots (separation). The wound will be primarily closed with individual sutures, and the sutures will be removed on the seventh postoperative day. After the surgical extraction of the third molar belonging the ozone therapy group, gaseous ozone will be applied to the extraction wound. Ozone will be reapplied 3 days after the intervention. After the surgical extraction of the third molar assigned to the sham ozone therapy, ozone will be applied by placing an inactive AV probe at the extraction site. The sham ozone therapy will also be applied 3 days after the surgical intervention. Postoperative instructions will be given to participants regarding oral hygiene maintenance, the use of cold compresses, and dietary recommendations. All participants will be invited for follow-up examinations on the 1st, 3rd and 7th day after the intervention.

Statistical data analysis will be conducted using SPSS version 20.0 (IBM SPSS Statistics for Windows, Version 20.0. Armonk, NY: IBM Corp, USA). Normality testing will be performed, and depending on the results, parametric and/or non-parametric tests will be applied. To compare differences between groups, chi-square tests, independent t-tests, and/or Mann-Whitney tests will be used. To determine differences within groups, paired t-tests and/or Wilcoxon tests will be applied. The correlation between variables will be determined using Pearson or Spearman correlation. A p-value of <0.05 will be considered statistically significant in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients with bilaterally impacted mandibular third molars classified as impaction index II B
* Patients in good general health (based on the ASA classification as ASA I and ASA II).

Exclusion Criteria:

* Contraindications for ozone application (pregnancy, hyperthyroidism, favism, anemia, myasthenia, bleeding disorders, alcohol intoxication, myocardial infarction, pacemaker, allergy to ozone)
* Patients who have used corticosteroid and antibiotic therapy in the last three months prior to inclusion in the study
* Patients with signs of local inflammation in the oral cavity
* Female patients during pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication: pain | 1st, 3rd, and 7th days after the intervention
  For the assessment of postoperative pain, the Numeric Visual Analogue Scale (VAS) (Carlsson, 1983) and the Verbal Rating Scale (VRS) (Aitken et al., 1969) will be used, which patients will complete. VAS is a horizontally drawn line of 100 mm in length, where the left end represents the absence of pain (0 mm), and the right end (100 mm) represents the worst pain ever experienced. The pain intensity will be determined by measuring the distance from the marked point on the scale to the left side of the scale and expressed in millimeters. The VRS is a numerical assessment of pain intensity based on six levels: 1 - no pain, 2 - very mild pain, 3 - mild pain, 4 - moderate pain, 5 - severe pain, 6 - very severe pain.
Postoperative complication: trismus | 1st, 3rd, and 7th days after the intervention
  The degree of postoperative trismus will be assessed by measuring the distance between the mesio-incisal angles of the upper and lower central incisors with the mouth fully open, using a caliper. The value will be expressed in millimeters (Marković and Todorović, 2007).
Postoperative complication: swelling | 1st, 3rd, and 7th days after the intervention
  The assessment of postoperative swelling will be performed by calculating the postoperative edema coefficient (Ec) using the modified formula by Carrillo et al. (1990): Postoperative distance - Preoperative distance x 100 /Preoperative distance. The postoperative Ec will be obtained by measuring in millimeters the preoperative and postoperative distances between the following reference points (R): AC - the most posterior point on the tragus to the lateral point at the corner of the mouth, AD - the most posterior point on the tragus to the prominent soft tissue landmark and BE - the lateral canthus of the eye to the lowest point on the angle of the mandible. Measurement will be done with a flexible ruler just before the intervention (the baseline value used for evaluating subsequent values).
Cytokine levels- wound healing | After surgical intervention, 3rd and 7th days after the intervention
  To determine the expression of IL-1β, IL-6, IL-8, TNF-α, VEGF, and TGF-β in samples from extraction wounds, real-time polymerase chain reaction (qPCR) will be used. Gene expression will be determined using "housekeeping" genes as standards and appropriate primers, according to the manufacturer's instructions. Each sample will be analyzed in duplicate.

SECONDARY OUTCOMES:
Quality of life | Before and on the 7th day after the intervention
  The Oral Health Impact Profile - 14 (Locker, 1998) will be used to assess quality of life. Possible The Oral Health Impact Profile - 14 scores range from 0 to 56, with higher score representing poor quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of East Sarajevo, Faculty of Medicine, Foča, Republika Srpska, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF
Time Frame: IPD supporting information will be available from January 2025 to the May 2025.
Access Criteria: Access to selected IPD (SAP, ICF) will have all researches from the principal investigator upon request.

REFERENCES:
- [Background] Markovic A, Todorovic Lj. Effectiveness of dexamethasone and low-power laser in minimizing oedema after third molar surgery: a clinical trial. Int J Oral Maxillofac Surg. 2007 Mar;36(3):226-9. doi: 10.1016/j.ijom.2006.10.006. Epub 2006 Dec 8. PMID 17157479
- [Background] Carrillo JS, Calatayud J, Manso FJ, Barberia E, Martinez JM, Donado M. A randomized double-blind clinical trial on the effectiveness of helium-neon laser in the prevention of pain, swelling and trismus after removal of impacted third molars. Int Dent J. 1990 Feb;40(1):31-6. PMID 2407660
- [Background] Aitken RC. Measurement of feelings using visual analogue scales. Proc R Soc Med. 1969 Oct;62(10):989-93. doi: 10.1177/003591576906201005. No abstract available. PMID 4899510
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] 34. Pell GJ, Gregory BT. Impacted mandibular third molars: Classification and Impacted mandibular third molars: Classification and modified technique for removal. Dent. Digest. 1933;39:330-8.